CLINICAL TRIAL: NCT04774796
Title: The Feasibility of a Group CBT Intervention for Improving Psychological Outcomes in Parents of Children With Food Allergy
Brief Title: Group CBT Intervention for Parents of Children With Food Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHMS 20-21 005 EGA
Record Dates: First submitted 2021-02-18; First posted 2021-03-01 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-08

CONDITIONS: Allergy;Food; Parents; Psychological Distress
MeSH Terms: conditions — Food Hypersensitivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental): Participants in this group will take part in a group CBT workshop for parents of children with food allergy. They will also have access to a self-help booklet in order to reinforce the learning that has taken place during the workshop.
  Interventions: Other: Cognitive Behavioural Therapy
- Treatment as usual (No Intervention): Participants in the control group will not take part in the group CBT workshop, but will have access to any treatment as usual relating to their child's food allergy. They will have access to the CBT self-help booklet after the all data collection has been finalised.

INTERVENTIONS:
Other: Cognitive Behavioural Therapy — Participants will take part in a one day, or two half-day group CBT workshop for parents of children with food allergy. The workshop will included understanding difficulties using a CBT model, psychoeducation on common psychological issues (e.g. anxiety) and the development of skills to help deal with maladaptive cognitions and behaviours relating to managing a child's food allergy.
  Arms: Cognitive Behavioural Therapy

SUMMARY:
Food allergy has been found to have a profound impact on parents of children with food allergy, with caregivers experiencing poorer psychological outcomes such as increased stress, anxiety, worry and depression than parents of non-allergic children. Furthermore, they report poorer quality of life (QoL) due to the psychosocial impact of looking after a child with food allergy, identifying the need for parental interventions aimed at improving these outcomes. There has generally been a paucity of research in this area, but there has recently been encouraging evidence to suggest that interventions involving Cognitive Behavioural Therapy (CBT) have the potential to improve the lives of those parents impacted by a child's food allergy. This study aims to add to this emerging evidence base by reporting on the feasibility of a brief, group CBT intervention for parents of children with food allergy. This small, proof of concept study also aims to report on a range of psychological measures to see if there is any evidence that this intervention may be effective in improving outcomes. Thirty to forty parents of children with food allergy will be recruited to the study and randomised to receive either a one-day or two half-day group CBT intervention or treatment as usual. Measures of a range of psychological outcomes, food allergy specific QoL and goal-based outcomes will be taken at baseline and at one and three-month follow ups. Participants will be asked for their feedback so that researchers can report on the acceptability of the intervention for those involved. This study is also interested in hearing about the parental experience of accessing psychological therapies as it is still not clear why some parents may require psychological intervention whilst others may not; participants in the intervention group will be invited to take part in interviews in order to share their experiences. It is hoped that this set of findings will help to determine if a brief group CBT intervention could be recommended for efficacy testing as part of a wider effort to provide evidence-based treatments for parents of children with food allergy experiencing poor psychological outcomes and poor food allergic-specific QoL.

DETAILED DESCRIPTION:
Food allergy is the adverse reaction of the body's immune system to the ingestion of food protein. When a food allergen is ingested, the immune system detects the food protein as a threat and releases a number of chemicals which cause the symptoms of an allergic reaction. These symptoms can include watery eyes, a running nose, itching, rashes, swelling and gastrointestinal problems, and may vary in their severity. Reactions can progress to anaphylaxis, which is a serious allergic reaction that is rapid in onset; symptoms can include a range of frightening respiratory, gastrointestinal and cardiovascular symptoms which may result in death if not treated promptly and effectively with adrenaline.

In the UK, food allergy is a prevalent problem, with an estimated 2 million people living with a diagnosed food allergy in the UK. Prevalence rates are higher in children than in adults, with an estimated 6-7% of children affected compared to 1-2% of adults, with this prevalence thought to be increasing. Currently, treatment involves avoidance of food allergens and the administration of treatment for accidently ingested foods.

The current management of food allergy involves the burden of constant vigilance, planning and preparation, with this responsibility often falling on parents (particularly the mothers) of young children. Furthermore, those with food allergy and their caregivers have to manage the unpredictable nature of food allergy and live continually with the risk and fear of accidental food ingestion which can negatively impact the Quality of Life (QoL) of allergy sufferers and their immediate family.

Research in this field has started to examine the psychological impact food allergy can not only have on the allergic child but also their parents. Previous studies have suggested that allergic children and their mothers experience higher stress and anxiety levels compared to the general population. Reasons why food allergy can cause such distress in parents include: the constant vigilance needed to check safety of foods; anxiety caused by severe and potentially fatal consequences of accidental ingestion of the food allergen; anxiety caused by handing over control of allergy management to the child (for example reading their own food labels); risk from the environment including people not understanding the impact of food allergy; worry about the future of their child, and dietary restrictions leading to social restrictions and potentially isolation. Given the impact looking after a child with food allergy can have on mental health and QoL in parents, the need for interventions to improve psychological outcomes is of high importance.

To date, there has been a paucity of research on interventions to improve psychological outcomes for parents of children with a food allergy. However, there is emerging evidence to suggest that Cognitive Behavioural Therapy (CBT) may be a promising intervention for parents experiencing poor psychological outcomes and QoL. CBT is a short-term therapy based on the rationale that what individuals think and do affects the way individuals feel. It has a strong evidence base for a range of mental health issues including anxiety and depression, and therefore may be appropriate for parents experiencing high levels of stress, anxiety and depression in relation to a child's food allergy. In the first study which reported on the effectiveness of CBT for mothers of children with a food allergy, five mothers received 12 weeks of individual face-to-face CBT, with six mothers acting as controls. All participants completed measures of anxiety, depression, worry, stress, general mental health, generic and food allergy specific QoL at baseline and at 12 weeks. Results showed that anxiety, depression and worry in the CBT group significantly reduced and overall mental health and QoL significantly improved from baseline to 12 weeks for mothers in the CBT group. A larger randomised control trial supported these promising initial findings. Two hundred mothers of children with food allergy were randomised to receive either a single-session CBT intervention or standard care, with anxiety and risk perception assessed at 6 weeks and 1 year. Results found significantly reduced state anxiety at six weeks in the intervention group, in the subgroup of mothers with moderate to high anxiety at enrolment and reduced risk perception. The study also found evidence of a reduction in physiological stress response in the intervention group, as measured by a salivary cortisol response to a simulated anaphylaxis scenario at one year. The results of both of these studies indicate that a CBT intervention may be an appropriate intervention for parents of children with food allergy.

This study seeks to add to this emerging evidence base by reporting on the feasibility of a brief group CBT intervention for improving psychological outcomes and food allergy specific QoL in parents of children with food allergy. There is already evidence that non-CBT-specific group interventions for parents with food allergic children can both be acceptable to parents and decrease parental burden, however, this study is the first to the researchers' knowledge to report on the feasibility of a brief group CBT intervention for parents of children with food allergy. Although a brief (one-day) intervention may seem optimistic in being able to bring about change, previous research in the field of child anxiety has shown promising evidence for the use of one-day interventions. A recent study has shown that children whose parents attended a one-day group intervention were 16.5% less likely to have an anxiety disorder than children whose parents received treatment as usual, highlighting than an inexpensive, one-day psycho-educational intervention may be useful in bringing about change. Group CBT interventions have the potential to offer a non-time consuming and cost-effective treatment option for parents of children with food allergy, an important factor for high in demand allergy services.

Qualitative research has provided insights into why food allergy can cause distress, however, reasons why parents access psychological support and their experiences of this, is still relatively unexplored. Differences in parental coping styles and levels of distress have been noted, indicating that only a sub-set of parents of food-allergic children may require psychological intervention. This study aims to speak to parents about their experiences of accessing psychological support (e.g. reasons for accessing psychological support, how other forms of support have helped/hindered and how they think a psychological intervention may help) in order to shed light on who CBT interventions may be most helpful for, and what CBT should comprise of for this group.

This study therefore is a contribution to the wider effort of providing evidence-based treatments for parents of children with food allergy impacted by the distressing psychosocial implications of caring for a food allergic child.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be the parent of at least one child with a diagnosed food allergy aged 0-17 years, currently experiencing difficulties with their wellbeing, in relation to their child's food allergy.

Exclusion Criteria:

* Individuals under the current care of a mental health care team or receiving any form of psychological intervention/treatment.
* Individuals taking part in another research study involving psychological intervention
* Individuals who do not have the capacity to provide informed consent
* Individuals who are not able to understand written and spoken English
* Individuals not able to access workshop materials (e.g. do not have an internet connection to take part in online workshops).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Food Allergy Quality of Life - Parental Burden Scale (Cohen et al., 2004) | Baseline, and 1 & 3 month follow ups
  17-item self-report scale which utilises a 7-point Likert scale in order to assess the burden of food allergy felt on the family. Higher scores represent greater parental burden.
Change in Depression, Anxiety and Stress Scales; short form version (Lovibond & Lovibond, 1995) | Baseline, and 1 & 3 month follow ups
  21-item self-report scale that is made up of three individual seven-item scales that measure depression, anxiety and stress. Higher scores represent higher levels of depression, anxiety and stress.
Change in Penn State Worry Questionnaire (Meyer et al., 1990) | Baseline, and 1 & 3 month follow ups
  16-item self-report scale to measure worry. Higher scores indicate greater worry.
Feedback questionnaire (researcher developed) | 3 month follow up
  Participants in the intervention group will be asked to complete a feedback questionnaire, in order for researchers to evaluate the CBT intervention and assess acceptability and feasibility.

SECONDARY OUTCOMES:
Change in Food Allergy Self-Efficacy Scale for Parents (Knibb, 2015) | Baseline, and 1 & 3 month follow ups
  21-item self-report scale with five subscales (managing social activities, precaution and prevention, allergic treatment, food allergen identification, and seeking information about food allergy). It is scored on a scale of 0-100, with higher scores indicate greater self-efficacy for food allergy management.
Change in Goal-Based Outcomes (researcher developed) | 1 & 3 month follow ups
  A goal-based outcome measure will be used to evaluate progress towards participant goals which will be collaboratively developed as part of the CBT intervention. This measure will be used for those in the intervention group only. Participants will be asked to rate the progress they feel they have made towards their goal from 0 to 10 (0 = no progress, 5 = exactly half-way to meeting the goal & 10 = met goal fully)

OTHER OUTCOMES:
Demographic Questionnaire (researcher developed) | Baseline
  A questionnaire to gather demographic information from the parent and food allergy information about their child.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Sherlock, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akeson N, Worth A, Sheikh A. The psychosocial impact of anaphylaxis on young people and their parents. Clin Exp Allergy. 2007 Aug;37(8):1213-20. doi: 10.1111/j.1365-2222.2007.02758.x. PMID 17651152
- [Background] Boyce JA, Assa'ad A, Burks AW, Jones SM, Sampson HA, Wood RA, Plaut M, Cooper SF, Fenton MJ, Arshad SH, Bahna SL, Beck LA, Byrd-Bredbenner C, Camargo CA Jr, Eichenfield L, Furuta GT, Hanifin JM, Jones C, Kraft M, Levy BD, Lieberman P, Luccioli S, McCall KM, Schneider LC, Simon RA, Simons FE, Teach SJ, Yawn BP, Schwaninger JM; NIAID-Sponsored Expert Panel. Guidelines for the Diagnosis and Management of Food Allergy in the United States: Summary of the NIAID-Sponsored Expert Panel Report. J Allergy Clin Immunol. 2010 Dec;126(6):1105-18. doi: 10.1016/j.jaci.2010.10.008. No abstract available. PMID 21134568
- [Background] Boyle RJ, Umasunthar T, Smith JG, Hanna H, Procktor A, Phillips K, Pinto C, Gore C, Cox HE, Warner JO, Vickers B, Hodes M. A brief psychological intervention for mothers of children with food allergy can change risk perception and reduce anxiety: Outcomes of a randomized controlled trial. Clin Exp Allergy. 2017 Oct;47(10):1309-1317. doi: 10.1111/cea.12981. Epub 2017 Aug 10. PMID 28710902
- [Background] Cartwright-Hatton S, Ewing D, Dash S, Hughes Z, Thompson EJ, Hazell CM, Field AP, Startup H. Preventing family transmission of anxiety: Feasibility RCT of a brief intervention for parents. Br J Clin Psychol. 2018 Sep;57(3):351-366. doi: 10.1111/bjc.12177. Epub 2018 Mar 25. PMID 29575043
- [Background] Cohen BL, Noone S, Munoz-Furlong A, Sicherer SH. Development of a questionnaire to measure quality of life in families with a child with food allergy. J Allergy Clin Immunol. 2004 Nov;114(5):1159-63. doi: 10.1016/j.jaci.2004.08.007. PMID 15536425
- [Background] Cummings AJ, Knibb RC, Erlewyn-Lajeunesse M, King RM, Roberts G, Lucas JS. Management of nut allergy influences quality of life and anxiety in children and their mothers. Pediatr Allergy Immunol. 2010 Jun;21(4 Pt 1):586-94. doi: 10.1111/j.1399-3038.2009.00975.x. Epub 2010 Jan 14. PMID 20088863
- [Background] Gillespie CA, Woodgate RL, Chalmers KI, Watson WT. "Living with risk": mothering a child with food-induced anaphylaxis. J Pediatr Nurs. 2007 Feb;22(1):30-42. doi: 10.1016/j.pedn.2006.05.007. PMID 17234496
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] King RM, Knibb RC, Hourihane JO. Impact of peanut allergy on quality of life, stress and anxiety in the family. Allergy. 2009 Mar;64(3):461-8. doi: 10.1111/j.1398-9995.2008.01843.x. Epub 2008 Dec 4. PMID 19076542
- [Background] Knibb RC. Effectiveness of Cognitive Behaviour Therapy for Mothers of Children with Food Allergy: A Case Series. Healthcare (Basel). 2015 Nov 25;3(4):1194-211. doi: 10.3390/healthcare3041194. PMID 27417820
- [Background] Knibb RC, Barnes C, Stalker C. Parental confidence in managing food allergy: development and validation of the Food Allergy Self-Efficacy Scale for Parents (FASE-P). Clin Exp Allergy. 2015 Nov;45(11):1681-9. doi: 10.1111/cea.12599. PMID 26215853
- [Background] Knibb RC, Semper H. Impact of suspected food allergy on emotional distress and family life of parents prior to allergy diagnosis. Pediatr Allergy Immunol. 2013 Dec;24(8):798-803. doi: 10.1111/pai.12176. PMID 24329879
- [Background] Knibb R, Halsey M, James P, du Toit G, Young J. Psychological services for food allergy: The unmet need for patients and families in the United Kingdom. Clin Exp Allergy. 2019 Nov;49(11):1390-1394. doi: 10.1111/cea.13488. Epub 2019 Sep 8. PMID 31454459
- [Background] Lau GY, Patel N, Umasunthar T, Gore C, Warner JO, Hanna H, Phillips K, Zaki AM, Hodes M, Boyle RJ. Anxiety and stress in mothers of food-allergic children. Pediatr Allergy Immunol. 2014 May;25(3):236-42. doi: 10.1111/pai.12233. PMID 24750570
- [Background] LeBovidge JS, Timmons K, Rich C, Rosenstock A, Fowler K, Strauch H, Kalish LA, Schneider LC. Evaluation of a group intervention for children with food allergy and their parents. Ann Allergy Asthma Immunol. 2008 Aug;101(2):160-5. doi: 10.1016/S1081-1206(10)60204-9. PMID 18727471
- [Background] Lopez-Lopez JA, Davies SR, Caldwell DM, Churchill R, Peters TJ, Tallon D, Dawson S, Wu Q, Li J, Taylor A, Lewis G, Kessler DS, Wiles N, Welton NJ. The process and delivery of CBT for depression in adults: a systematic review and network meta-analysis. Psychol Med. 2019 Sep;49(12):1937-1947. doi: 10.1017/S003329171900120X. Epub 2019 Jun 10. PMID 31179960
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Roy KM, Roberts MC. Peanut allergy in children: relationships to health-related quality of life, anxiety, and parental stress. Clin Pediatr (Phila). 2011 Nov;50(11):1045-51. doi: 10.1177/0009922811412584. Epub 2011 Jun 17. PMID 21685213
- [Background] Sicherer SH, Sampson HA. Food allergy. J Allergy Clin Immunol. 2010 Feb;125(2 Suppl 2):S116-25. doi: 10.1016/j.jaci.2009.08.028. Epub 2009 Dec 29. PMID 20042231
- [Background] Sugunasingha N, Jones FW, Jones CJ. Interventions for caregivers of children with food allergy: A systematic review. Pediatr Allergy Immunol. 2020 Oct;31(7):805-812. doi: 10.1111/pai.13255. Epub 2020 Jun 24. PMID 32311157
- [Background] Turner PJ, Gowland MH, Sharma V, Ierodiakonou D, Harper N, Garcez T, Pumphrey R, Boyle RJ. Increase in anaphylaxis-related hospitalizations but no increase in fatalities: an analysis of United Kingdom national anaphylaxis data, 1992-2012. J Allergy Clin Immunol. 2015 Apr;135(4):956-963.e1. doi: 10.1016/j.jaci.2014.10.021. Epub 2014 Nov 25. PMID 25468198
- [Background] Valentine AZ, Knibb RC. Exploring quality of life in families of children living with and without a severe food allergy. Appetite. 2011 Oct;57(2):467-74. doi: 10.1016/j.appet.2011.06.007. Epub 2011 Jun 25. PMID 21708202
- [Background] van Dis EAM, van Veen SC, Hagenaars MA, Batelaan NM, Bockting CLH, van den Heuvel RM, Cuijpers P, Engelhard IM. Long-term Outcomes of Cognitive Behavioral Therapy for Anxiety-Related Disorders: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2020 Mar 1;77(3):265-273. doi: 10.1001/jamapsychiatry.2019.3986. PMID 31758858
- [Derived] Jones CJ, Tallentire H, Edgecumbe R, Sherlock G, Hale L. Online, group, low-intensity psychological intervention for adults, children, and parents with food allergy. Ann Allergy Asthma Immunol. 2024 Oct;133(4):453-461. doi: 10.1016/j.anai.2024.07.025. Epub 2024 Jul 26. PMID 39069154
- See also: The Natasha Allergy Research Foundation (2019). The Allergy Explosion. Retrieved from https://www.narf.org.uk/the-allergy-explosion. — https://www.narf.org.uk/the-allergy-explosion